CLINICAL TRIAL: NCT02161224
Title: A Phase 1, Non-randomized, Open-label, Single-dose Study to Investigate the Pharmacokinetics, Safety and Tolerability of FG-4592 in Subjects With Moderate Hepatic Impairment and Healthy Subjects With Normal Hepatic Function
Brief Title: A Study to Investigate the Exposure and Safety and Tolerability of a Single Dose of FG-4592 in Subjects With Moderately Diminished Liver Function Compared to Those With Normal Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1517-CL-0513; 2013-001533-41 (EudraCT Number)
Record Dates: First submitted 2014-06-09; First posted 2014-06-11 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: PK of FG-4592; Hepatic Insufficiency; Healthy Subjects
Keywords: Phase 1; FG-4592; Single dose; Moderate hepatic impairment
MeSH Terms: conditions — Hepatic Insufficiency | interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: FG-4592 in subjects with moderate hepatic impairment (Experimental)
  Interventions: Drug: FG-4592
- 2: FG-4592 in healthy subjects (Experimental)
  Interventions: Drug: FG-4592

INTERVENTIONS:
Drug: FG-4592 — Oral
  Other Names: ASP1517,; roxadustat

SUMMARY:
The effect of moderately diminished liver function on the exposure, safety and tolerability of a single dose of FG-4592 is studied in male and female subjects. The results are compared to the data gained from subjects with normal liver function.

DETAILED DESCRIPTION:
The effect of moderate hepatic impairment on the pharmacokinetics (PK), safety and tolerability of a single dose of FG-4592 in male and female subjects is investigated. Data obtained from these subjects are compared to data from BMI-, age- and sex-matched subjects with normal hepatic function. Both groups consist of 8 subjects.

Screening takes place from Days -22 to -2 before admission to the clinical unit on Day -1. Administration of the trial medication takes place on Day 1 under fasted conditions. Healthy subjects are discharged on Day 5 and subjects with moderate hepatic impairment on Day 7, if there is no reason to extend the stay. An end-of-study visit (ESV) takes place 5 to 9 days after (early) discharge.

Safety assessments are performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Both healthy subjects and subjects with moderate hepatic impairment:

* Independent Ethics Committee (IEC)-approved written Informed Consent and privacy language as per national regulations must be obtained from the subject prior to any study-related procedures (including withdrawal of prohibited medication, if applicable).
* Male subjects and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening and continuing throughout the study period and for 90 days after the study drug administration.

In addition, subjects with moderate hepatic impairment must also meet the following inclusion criteria:

* Subject has Child-Pugh classification Class B (moderate, 7 to 9 points) liver function impairment [screening].

Exclusion Criteria:

Both healthy subjects and subjects with moderate hepatic impairment:

* Female subject who has been pregnant within 6 months prior to screening or breastfeeding within 3 months before screening.
* Subject has a known or suspected hypersensitivity to FG-4592, or any components of the formulation used.

In addition, healthy subjects must also NOT meet the following exclusion criteria:

* Subject has any of the liver function tests (LFT) (Aspartate Aminotransferase [AST], Alanine Aminotransferase [ALT], Alkaline Phosphatase [ALP], Gamma Glutamyl Transferase [GGT], Total Bilirubin [TBL] above the upper limit of normal (ULN). In such a case the assessment may be repeated once [Day-1].

In addition, subjects with moderate hepatic impairment must also NOT meet the following exclusion criteria:

* Subject had a previous liver transplantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of FG-4592 in plasma as measured by area under the concentration-time curve (AUC) extrapolated to infinity (AUCinf) | Days 1 to 5 (Day 7 for hepatic impaired subjects)
Pharmacokinetic parameter of FG-4592 in plasma as measured by maximum concentration (Cmax) | Days 1 to 5 (Day 7 for hepatic impaired subjects)

SECONDARY OUTCOMES:
Pharmacokinetic profile of FG-4592 in plasma | Days 1 to 5 (Day 7 for hepatic impaired subjects)
  AUC up to last quantifiable concentration (AUClast), AUC from 0 up to last quantifiable concentration based on unbound plasma concentration (AUClast,u), AUC from time point 0 to time point 24 hours (AUC0-24h), AUC from time point 0 to time point 24 hours based on unbound plasma concentration (AUC0-24h,u), unbound AUC extrapolated to infinity (AUCinf,u), unbound maximum concentration (observed) (Cmax,u), apparent total systemic clearance after extra-vascular dosing (CL/F), plasma clearance over bioavailability ratio based on unbound plasma (CLu/F), fraction unbound (fu), lag-time (time delay between drug administration and first observed concentration above the Limit of Quantification (LOQ) in plasma) (tlag), time to attain Cmax (tmax), apparent terminal elimination half-life (t1/2), apparent volume of distribution during terminal phase after oral administration (Vz/F), unbound apparent volume of distribution during terminal phase after oral administration (Vz,u/F)
Pharmacokinetic profile of FG-4592 in urine | Days 1 to 5 (Day 7 for hepatic impaired subjects)
  renal clearance (CLR), renal clearance based on unbound concentration (CLR,u), renal clearance from time point 0 to 24 hours (CLR,0-24h), renal clearance from time point 0 to 24 hours based on unbound concentration (CLR,u 0-24h), amount of unchanged drug excreted into urine from time point 0 to infinity (Aeinf), amount of unchanged drug excreted into urine from time point 0 to infinity, percentage of dose (Aeinf%), amount of unchanged drug excreted into urine until the last observation time point (Aelast), amount of unchanged drug excreted into urine until the last observation time, percentage of dose (Aelast%), amount of drug excreted into urine from time point 0 to time point 24 hours (Ae0-24h), amount of drug excreted into urine from time point 0 to time point 24 hours, percentage of dose (Ae0-24h%)
Erythropoietin in plasma | Days 1 to 5 (Day 7 for hepatic impaired subjects)
  maximum achievable pharmacologic effect (Emax), area under the concentration-time curve from 0 up to last quantifiable concentration based on EPO concentration (AUCE,last), tmax
Safety and tolerability of FG-4592 | Screening (Days -22 to -2) to ESV (5 to 9 days after (early) discharge)
  Nature, frequency and severity of adverse events (AEs), vital signs, safety laboratory tests, electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Central contact, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- COMAC, Sofia, Bulgaria